CLINICAL TRIAL: NCT00585936
Title: Evaluation of Magnetic Nanoparticle Enhanced Imaging in Autoimmune Diabetes
Brief Title: Imaging Inflammation in Autoimmune Diabetes
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Massachusetts General Hospital (Other); AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Joslin 06-32; P01-A1-054904
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Normal controls without evidence of diabetes or islet specific autoimmunity
- 2: Individuals within 6 months of diagnosis with type 1 diabetes
- 3: Individuals at high risk for the development of type 1 diabetes
- 4: Individuals with longstanding autoimmune diabetes

SUMMARY:
The purpose of this study is to determine whether magnetic resonance imaging (MRI) with ferumoxtran-10 can be used to detect changes in the pancreas associated with autoimmune diabetes.

DETAILED DESCRIPTION:
Approximately one million individuals are afflicted with autoimmune Type 1 diabetes mellitus (T1DM) in the United States. This disease results from the autoimmune destruction of the insulin-producing beta-cells of the islets of Langerhans of the pancreas. Initially, diabetes is usually clinically occult with localized pancreatic inflammation characterized by a lymphocytic infiltration of the pancreatic islets, termed insulitis, which leads to beta-cell specific destruction of the islets. This is often followed by the clinically overt phase that ensues when the bulk of beta cells have been destroyed and the pancreas is no longer able to produce sufficient insulin to maintain glycemic control. The purpose of this study is to assess the ability of magnetic resonance imaging with ferumoxtran-10, a functional molecular imaging agent consisting of iron oxide nanoparticles, to detect changes in the pancreas associated with the insulitis of T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Recent onset type 1 diabetes as defined by clinical diagnosis within the last 6 months and age less than 30 or at least one islet autoantibody marker (GAD, IAA, or IA-2).

or

* High risk of pre-type 1 diabetes as defined by first degree family relative with type 1 diabetes and at least one islet autoantibody marker (GAD, IAA, or IA-2).

or

* Individuals with established type 1 diabetes of greater than 6 months duration who were under age 30 or at least one islet autoantibody marker positive (GAD, IAA, or IA-2) at time of diagnosis or who currently are GAD or IA-2 autoantibody marker positive.

or

* Normal control as defined by no family history of type 1 diabetes and normal tolerance test (tolerance testing to be performed as part of protocol).

Exclusion Criteria:

* Individuals under 18 years of age
* Individuals unable or unwilling to give informed consent/HIPAA authorization
* Individuals who are clinically unstable
* Individuals with any contraindications to MRI examination, for example, individuals with pacemakers
* Pregnant or lactating women
* Individuals with allergies to iron or dextran
* Individuals with a history of cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is to be drawn from the general population, diabetes clinic population, and at risk individuals as previously identified in prior family studies.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Jackson, M.D., Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Turvey SE, Swart E, Denis MC, Mahmood U, Benoist C, Weissleder R, Mathis D. Noninvasive imaging of pancreatic inflammation and its reversal in type 1 diabetes. J Clin Invest. 2005 Sep;115(9):2454-61. doi: 10.1172/JCI25048. Epub 2005 Aug 18. PMID 16110329
- [Background] Denis MC, Mahmood U, Benoist C, Mathis D, Weissleder R. Imaging inflammation of the pancreatic islets in type 1 diabetes. Proc Natl Acad Sci U S A. 2004 Aug 24;101(34):12634-9. doi: 10.1073/pnas.0404307101. Epub 2004 Aug 10. PMID 15304647
- [Result] Gaglia JL, Guimaraes AR, Harisinghani M, Turvey SE, Jackson R, Benoist C, Mathis D, Weissleder R. Noninvasive imaging of pancreatic islet inflammation in type 1A diabetes patients. J Clin Invest. 2011 Jan;121(1):442-5. doi: 10.1172/JCI44339. Epub 2010 Dec 1. PMID 21123946